CLINICAL TRIAL: NCT03701399
Title: A Phase III, Long-Term, Randomized, Double-blind, Placebo-controlled Trial of Troriluzole in Adult Participants With Spinocerebellar Ataxia.
Brief Title: Troriluzole in Adult Participants With Spinocerebellar Ataxia
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biohaven Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BHV4157-206
Expanded Access: NCT06034886 (Available)
Record Dates: First submitted 2018-10-05; First posted 2018-10-10 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Spinocerebellar Ataxias; Spinocerebellar Ataxia Type 1; Spinocerebellar Ataxia Type 2; Spinocerebellar Ataxia Type 3; Spinocerebellar Ataxia Type 6; Spinocerebellar Ataxia Type 7; Spinocerebellar Ataxia Type 8; Spinocerebellar Ataxia Type 10
Keywords: Ataxia, SCA, Spinocerebellar Ataxia
MeSH Terms: conditions — Spinocerebellar Ataxias; Machado-Joseph Disease; Spinocerebellar ataxia 8; Spinocerebellar Ataxia 10; Ataxia; Heart Arrest

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Troriluzole (Experimental): Randomization phase (Randomization through Week 48):
  Participants received starting dose of troriluzole 140 milligrams (mg) capsules orally once daily for first 4 weeks, followed by 200 mg once daily for the remaining 44 weeks of 48-week duration of the double-blind randomization phase.
  Open-label extension (OLE) phase (OLE Week 1 up to Week 192): Participants who were eligible and agreed to enroll in an OLE phase, will receive troriluzole 200 mg capsules orally once daily for 4 weeks in a blinded manner. After OLE Week 4, all participants will then receive open label troriluzole 200 mg up to Week 192.
  Interventions: Drug: troriluzole
- Placebo (Placebo Comparator): Randomization phase (Randomization through Week 48):
  Participants received troriluzole matching placebo capsules orally once daily for 48 weeks duration of the double-blind randomization phase.
  OLE phase (Week 1 up to Week 192): Participants who were eligible and agreed to enroll in an OLE phase, will receive troriluzole 140 mg capsules orally once daily for the first 4 weeks in a blinded manner. After OLE Week 4, all participants will then receive open label troriluzole 200 mg up to Week 192.
  Interventions: Drug: troriluzole; Drug: Placebo

INTERVENTIONS:
Drug: troriluzole — Administered orally
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the efficacy of Troriluzole (200 mg once daily) versus placebo after 48 weeks of treatment in subjects with spinocerebellar ataxia (SCA).

ELIGIBILITY:
Inclusion Criteria:

1. Participants with a known or suspected diagnosis of the following specific hereditary ataxias: SCA1, SCA2, SCA3, SCA6, SCA7, SCA8 and SCA10.

   1. A participant should have a confirmed genotypic diagnosis from a Clinical Laboratory Improvement Amendments (CLIA) certified lab (can produce test results); or,
   2. A participant has a family member that has a confirmed genotypic diagnosis from a CLIA certified lab (can produce test results) and must be willing to undergo genetic testing to confirm underlying SCA diagnosis; or,
   3. A participant has a confirmed genotypic diagnosis from a lab that is not CLIA certified and must be willing to undergo genetic testing to confirm underlying SCA diagnosis; or,
   4. A participant has clinical evidence that supports diagnosis of one of the aforementioned SCA genotypes but does not have producible test results from a CLIA certified lab from either a family member or for his or herself and the participant must be willing to undergo such testing to confirm the SCA diagnosis (in this case, site must wait for results of genotypic testing prior to randomization)
2. Ability to ambulate 8 meters without human assistance (canes and other devices allowed)
3. Screening Modified Functional Scale for the Assessment and Rating of Ataxia (f-SARA) total score ≥3.
4. Score of ≥1 on gait subsection of the f-SARA
5. Determined by the investigator to be medically stable at Baseline/randomization as assessed by medical history, physical examination, laboratory test results, and electrocardiogram testing.

Exclusion Criteria:

1. A ≥ 2-point difference on the Modified Functional SARA score between screening and baseline
2. Mini Mental State Exam (MMSE) score <24
3. Any medical condition other than one of the hereditary ataxias specified in the inclusion criteria that could predominantly explain or contribute significantly to the participants' symptoms of ataxia.
4. A prominent spasticity or dystonia that, in the opinion of the investigator, will compromise the ability of the SARA instrument to assess underlying ataxia severity.
5. A score of 4 on any individual item (Items 1-4) of the f-SARA
6. Participants should be excluded at screening or baseline if medical conditions have arisen or there is a change in disease status that could confound the ability of the SARA to accurately reflect changes in ataxia severity.
7. Active liver disease or a history of hepatic intolerance to medications that in the investigator's judgment, is medically significant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2026-06 (Estimated)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (21):
  - Barrow Neurological Institute, Phoenix, Arizona
  - CNS Trials, Long Beach, California
  - UCLA, Los Angeles, California
  - UCSF, San Francisco, California
  - University of Colorado Hospital, Aurora, Colorado
  - University of Florida Health, Gainesville, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - University of South Florida, Tampa, Florida
  - Emory, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Northwest Neurology, Ltd., Rolling Meadows, Illinois
  - Johns Hopkins Medicine, Lutherville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Columbia University, New York, New York
  - Duke University Movement Disorders Clinic, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Houston Methodist, Houston, Texas
  - Swedish Health Services, Seattle, Washington
- China (2):
  - Central South University Xiangya Hospital, Changsha, Hunan
  - West China Hospital of Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Potashman MH, Popoff E, Powell LC, Beiner MW, Mackenzie A, Coric V, Subramony S, Synofzik M, Schmahmann J, L'Italien G. Measurement Properties of the Friedreich Ataxia Rating Scale in Patients with Spinocerebellar Ataxia. Neurol Ther. 2025 Apr;14(2):527-545. doi: 10.1007/s40120-024-00708-4. Epub 2025 Jan 13. PMID 39806095
- [Derived] L'Italien GJ, Oikonomou EK, Khera R, Potashman MH, Beiner MW, Maclaine GDH, Schmahmann JD, Perlman S, Coric V. Video-Based Kinematic Analysis of Movement Quality in a Phase 3 Clinical Trial of Troriluzole in Adults with Spinocerebellar Ataxia: A Post Hoc Analysis. Neurol Ther. 2024 Aug;13(4):1287-1301. doi: 10.1007/s40120-024-00625-6. Epub 2024 May 30. PMID 38814532
- [Derived] Schmahmann JD, Pierce S, MacMore J, L'Italien GJ. Development and Validation of a Patient-Reported Outcome Measure of Ataxia. Mov Disord. 2021 Oct;36(10):2367-2377. doi: 10.1002/mds.28670. Epub 2021 Jun 11. PMID 34115419

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 23 sites in 2 countries (21 sites in the US and 2 sites in China).
Pre-assignment Details: A total of 299 participants were enrolled, of which 218 participants were randomized in a 1:1: ratio to receive troriluzole or placebo. Study consisted of double-blind randomization phase (up to Week 48) and open-label extension phase (up to Week 192). The study is ongoing, and results are reported only for randomization phase (up to Week 48).
Groups:
- Troriluzole: Randomization phase (Randomization through Week 48):
  Participants received starting dose of troriluzole 140 milligrams (mg) capsules orally once daily for first 4 weeks, followed by 200 mg once daily for the remaining 44 weeks of 48 week duration of the double-blind randomization phase.
  Open-label extension (OLE) phase (OLE Week 1 up to Week 192): Participants who were eligible and agreed to enroll in an OLE phase, will receive troriluzole 200 mg capsules orally once daily for 4 weeks in a blinded manner. After OLE Week 4, all participants will then receive open label troriluzole 200 mg up to Week 192.
Period: Overall Study
Arm/Group | Troriluzole | Placebo
Started | 109 | 109
Treated | 108 | 109
Completed | 96 | 96
Not Completed | 13 | 13
Not completed — Adverse Event | 3 | 5
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Investigators decision | 1 | 2
Not completed — Lost to Follow-up | 1 | 2
Not completed — Death | 1 | 1
Not completed — Randomized but not treated | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated analysis set (TAS): The treated analysis set included all randomized/enrolled participants who received at least one dose of study medication (blinded or open label troriluzole, or blinded placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | Troriluzole | Placebo | Total
Number analyzed (Participants) | 108 | 109 | 217
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (13.16) | 47.6 (12.48) | 47.6 (12.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 56 | 106
  Male | 58 | 53 | 111
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 11 | 24
  Not Hispanic or Latino | 95 | 98 | 193
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 19 | 21 | 40
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 14 | 26
  White | 74 | 74 | 148
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Number of Participants with Spinocerebellar ataxia (SCA) Genotype [Number; unit: participants]
  SCA1 | 15 | 11 | 26
  SCA2 | 32 | 35 | 67
  SCA3 | 44 | 45 | 89
  SCA6 | 6 | 6 | 12
  SCA7 | 5 | 5 | 10
  SCA8 | 3 | 2 | 5
  SCA10 | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Randomization Phase: Change From Baseline in the Modified Functional Scale for the Assessment and Rating of Ataxia (f-SARA) Total Score at Week 48 in SCA Participants
Description: The f-SARA was a 4-item performance based scale: 1-gait, 2-stance, 3-sitting, 4-speech disturbance (0:normal (no impairment), 1: mildly impaired function, but no assistance required, 2: moderately impaired function, but needs assistance for certain parts of task, 3: severely impaired function to degree that assistance is needed for all parts of the task, 4: unable to perform function). Total score was derived as sum of individual items; ranged from 0 to 16. Higher score indicated worst outcome. A negative change in score showed improvement.
Time Frame: Randomization Baseline; Week 48
Population: The modified intent-to-treat (mITT) analysis set in randomization phase included randomized participants who received at least one dose of double-blind study medication (troriluzole or placebo) during the randomization phase and provided a non-missing baseline measurement and at least one non-missing post-baseline efficacy measurement during the randomization phase. Participants with available data were included. Pre-specified randomization strata by SCA genotype.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Troriluzole: Randomization phase (Randomization through Week 48):
  Participants received starting dose of troriluzole 140 milligrams (mg) capsules orally once daily for first 4 weeks, followed by 200 mg once daily for the remaining 44 weeks of 48 week duration of the double-blind randomization phase.
- Placebo: Randomization phase (Randomization through Week 48):
  Participants received troriluzole matching placebo capsules orally once daily for 48 weeks duration of the double-blind randomization phase.
Arm/Group | Troriluzole | Placebo
Number analyzed (Participants) | 94 | 95
score on a scale
  All SCA | 0.20 (0.19) | 0.27 (0.18)
  SCA3: number analyzed (Participants) | 38 | 40
  SCA3 | -0.03 (0.20) | 0.53 (0.19)
Statistical Analysis 1: Comparison: Troriluzole vs Placebo; All SCA participants; Test type: Superiority; p = 0.7581, Mixed Models Analysis; Least squares mean difference = -0.06, 95% CI 2-sided [-0.47 to 0.34], Standard Error of Mean 0.20 — Model based summary statistics were from a mixed model with repeated measures, including fixed effects for treatment, randomization stratum (SCA genotype group), visit, treatment-by-visit interaction, and country, baseline score as a covariate
Statistical Analysis 2: Comparison: Troriluzole vs Placebo; SCA3 genotype participants; Test type: Superiority; p = 0.0450, Mixed Models Analysis; Least square mean difference = -0.56, 95% CI 2-sided [-1.11 to -0.01], Standard Error of Mean 0.28 — Model based summary statistics were from a mixed model with repeated measures, including fixed effects for treatment, randomization stratum (SCA genotype group), visit, treatment-by-visit interaction, and country

2. Secondary Outcome: Randomization Phase: Change From Baseline in Patient Impression of Function and Activities of Daily Living Scale (PIFAS) Total Score at Week 48 in SCA Participants
Description: PIFAS was a 17-item instrument designed to assess the level of functional disability. The scale was rater administered and the items were selected to encompass domains of relevance to SCA (i.e., mobility, speech/swallowing, and fatigue), and to capture function and activities of daily living within these domains. Statements were rated on a 5-point Likert scale ranging from "0" reflecting "not at all" to "4" reflecting "very much." The total score was derived as the sum of the individual items, ranged between 0 to 68. Higher score indicated a worst outcome. A negative change in score showed improvement.
Time Frame: Randomization Baseline, Week 48
Population: Participants in mITT analysis set with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Troriluzole | Placebo
Number analyzed (Participants) | 94 | 90
score on a scale
  All SCA | -0.93 (1.49) | 1.03 (1.43)
  SCA3: number analyzed (Participants) | 38 | 37
  SCA3 | 0.56 (1.65) | 2.96 (1.67)

3. Secondary Outcome: Randomization Phase: Change From Baseline in Friedreich's Ataxia Rating Scale - Activities of Daily Living (FARS-ADL) Total Score at Week 48 in SCA Participants
Description: FARS was a scale consisting of combined timed measures of performance, FUNC (0-6, higher score indicated worst outcome), ADL with paramount neurologic examination (0-36, higher score indicated worst outcome), FARSn (0-125, higher score indicated worst outcome). Total score was sum of these 3 subscales: 0-167, higher score indicated worst outcome. For this outcome measure, only FARS-ADL sub-scale was evaluated. It was multicomponent scale designed to assess neurological domains affected in Friedreich's Ataxia, another hereditary cerebellar ataxia disorder. This subscale had been validated in Friedreich's ataxia, was a measure of functional disability, and correlated with SARA total scores. It assessed 9 areas of ADL with response categories rated on 5-point scale with "0" reflecting "normal" and "4" reflecting inability to perform specific function. Total score was derived as sum of individual items, ranging 0-36, higher score indicated worst outcome. FARS-ADL was rater administered.
Time Frame: Randomization Baseline, Week 48
Population: Participants in mITT analysis set with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Troriluzole | Placebo
Number analyzed (Participants) | 94 | 95
score on a scale
  All SCA | 0.453 (0.502) | -0.017 (0.480)
  SCA3: number analyzed (Participants) | 37 | 39
  SCA3 | 0.918 (0.523) | 1.130 (0.506)

4. Secondary Outcome: Randomization Phase: Change From Baseline in Functional Staging for Ataxia Scale From the Friedreich's Ataxia Rating Scale (FARS-FUNC) Total Score at Week 48 in SCA Participants
Description: FARS was a scale consisting of combined timed measures of performance, FUNC (0-6, higher score indicated worst outcome), ADL with paramount neurologic examination (0-36, higher score indicated worst outcome), FARSn (0-125, higher score indicated worst outcome). The total score was a sum of these 3 subscales; 0-167, higher score indicated worst outcome.
  For this outcome measure, only the FARS-FUNC sub-scale was evaluated. FARS-FUNC was a subscale of the FARS designed to provide functional staging for ataxia in which clinicians were asked to assess function on a 6-stage staging system, with "0" reflecting "normal" and "6" reflecting a stage in participant was "total disabled".
Time Frame: Randomization Baseline, Week 48
Population: Participants in mITT analysis set with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Placebo: Participants received troriluzole matching placebo capsules orally once daily for 48 weeks duration of the double-blind randomization phase.
Arm/Group | Troriluzole | Placebo
Number analyzed (Participants) | 93 | 94
score on a scale
  All SCA | 0.266 (0.075) | 0.226 (0.072)
  SCA3: number analyzed (Participants) | 37 | 39
  SCA3 | 0.216 (0.079) | 0.328 (0.077)

5. Secondary Outcome: Randomization Phase: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Serious Adverse Events (TESAEs); and AEs Leading to Treatment Discontinuation
Description: An AE was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a participant that did not necessarily had a causal relationship with this treatment. An SAE was defined as any AE that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect in the offspring of the participant or was considered another important medical event. Treatment-emergent AEs (TEAEs) in the randomization phase included any AE with an onset date on or after the first day of double-blind study drug and up to the first day of open-label study drug in the extension phase (for participants entering the extension phase) or last day of the randomization phase study drug + 30 days.
Time Frame: From first dose of study drug to Week 48 plus 30 days (maximum duration: 52 weeks)
Population: The treated analysis set (TAS) included all randomized/enrolled participants who received at least one dose of study medication (blinded or open label troriluzole, or blinded placebo).
Measure: Number; unit: participants
Groups:
- Placebo: Randomization phase (Randomization through Week 48):
  Participants received troriluzole matching placebo capsules orally once daily for 48 weeks duration of the double-blind randomization phase.
  .
Arm/Group | Troriluzole | Placebo
Number analyzed (Participants) | 108 | 109
participants
  TEAEs | 87 | 92
  TESAEs | 6 | 8
  AEs Leading to Treatment Discontinuation | 5 | 5

6. Other Pre Specified Outcome: Randomization Phase: Change From Baseline in the f-SARA Total Score at Week 48 in SCA3 Participants
Description: The f-SARA was a 4-item performance based scale: 1-gait, 2-stance, 3-sitting, 4-speech disturbance (0:normal (no impairment), 1:mildly impaired function, but no assistance required, 2:moderately impaired function, but needs assistance for certain parts of task, 3: severely impaired function to degree that assistance is needed for all parts of the task, 4:unable to perform function). Total score was derived as sum of individual items; ranged from 0 to 16. Higher score indicated worst outcome. A negative change in score shows improvement.
Time Frame: Randomization Baseline; Week 48
Population: Participants in mITT analysis set with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Troriluzole | Placebo
Number analyzed (Participants) | 38 | 40
score on a scale | -0.03 (0.20) | 0.53 (0.19)

7. Other Pre Specified Outcome: Randomization Phase: Change From Baseline in PIFAS Total Score at Week 48 in SCA3 Participants
Description: PIFAS was a 17-item instrument designed to assess the level of functional disability. The scale is rater administered and the items were selected to encompass domains of relevance to SCA (i.e., mobility, speech/swallowing, and fatigue), and to capture function and activities of daily living within these domains. Statements are rated on a 5-point Likert scale ranging from "0" reflecting "not at all" to "4" reflecting "very much." The total score is derived as the sum of the individual items, ranged between 0 to 68. Higher score indicated a worst outcome. A negative change in score showed improvement.
Time Frame: Randomization Baseline, Week 48
Population: Participants in mITT analysis set with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Troriluzole | Placebo
Number analyzed (Participants) | 38 | 37
score on a scale | 0.56 (1.65) | 2.96 (1.67)

8. Other Pre Specified Outcome: Randomization Phase: Change From Baseline in FARS-ADL Total Score at Week 48 in SCA3 Participants
Description: as for outcome 3
Time Frame: Randomization Baseline, Week 48
Population: Participants in mITT analysis set with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Troriluzole | Placebo
Number analyzed (Participants) | 37 | 39
score on a scale | 0.918 (0.523) | 1.130 (0.506)

9. Other Pre Specified Outcome: Randomization Phase: Change From Baseline in FARS-FUNC Total Score at Week 48 in SCA3 Participants
Description: as for outcome 4
Time Frame: Randomization Baseline, Week 48
Population: Participants in mITT analysis set with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Troriluzole | Placebo
Number analyzed (Participants) | 37 | 39
score on a scale | 0.216 (0.079) | 0.328 (0.077)

10. Other Pre Specified Outcome: Change From Baseline in Clinical Global Impression - Global Improvement Scale (CGI-I) in SCA3 Participants
Description: The CGI-I was a 7-point scale that required the clinician to assess how much the participant's illness had improved or worsened relative to the baseline visit and it was rated on a 7 point scale: 1= "Very much improved", 2= "Much improved", 3= "Minimally improved", 4= "No change", 5= "Minimally worse", 6= "Much worse" and 7= "Very much worse". Higher scores indicated greater impairment.
Time Frame: Randomization Baseline; Week 48
Population: Participants in mITT analysis set with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Troriluzole | Placebo
Number analyzed (Participants) | 35 | 38
score on a scale | 4.14 (0.17) | 4.68 (0.17)

11. Other Pre Specified Outcome: Falls Events in Troriluzole Compared to Placebo for All SCA Participants
Description: An AE of Fall was recorded if there was a worsening of frequency of falls or if a fall was associated with an injury.
Time Frame: Randomization Baseline, Week 48
Population: All randomized participants who received at least one dose of study medication during the randomization phase.
Measure: Number; unit: Number of events
Groups:
- Troriluzole: Randomization phase (Randomization through Week 48) Participants received starting dose of troriluzole 140 milligrams (mg) capsules orally once daily for first 4 weeks, followed by 200 mg once daily for the remaining 44 weeks of 48-week duration of the double-blind randomization phase.
- Placebo: Randomization phase (Randomization through Week 48) Participants received troriluzole matching placebo capsules orally once daily for 48 weeks duration of the double-blind randomization phase.
Arm/Group | Troriluzole | Placebo
Number analyzed (Participants) | 108 | 109
Number of events | 20 | 42

ADVERSE EVENTS:
Time Frame: For Adverse events (AEs): From first dose of study drug up to Week 48 plus 30 days (maximum duration: 52 weeks) For All-cause mortality: From randomization up to Week 48 plus 30 days (maximum duration: 52 weeks)
Description: For AEs: The treated analysis set (TAS) included all randomized/enrolled participants who received at least one dose of study medication (blinded or open label troriluzole, or blinded placebo)
  For All-cause mortality: All randomized participants.
Arm/Group | Troriluzole | Placebo
All-Cause Mortality (participants affected / at risk) | 1/109 | 1/109
Serious Adverse Events (participants affected / at risk) | 6/108 | 8/109
Other Adverse Events (participants affected / at risk) | 54/108 | 58/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Troriluzole (N=108) | Placebo (N=109)
Fall (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Pulmonary contusion (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Human chorionic gonadotropin positive (Investigations) | 1 | 0
Liver function test increased (Investigations) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 2
Abscess (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Pneumatosis (General disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Haematocoele (Vascular disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 2
Major depression (Psychiatric disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Troriluzole (N=108) | Placebo (N=109)
Headache (Nervous system disorders) | 13 | 8
Dizziness (Nervous system disorders) | 9 | 11
Fall (Injury, poisoning and procedural complications) | 13 | 24
Contusion (Injury, poisoning and procedural complications) | 7 | 7
Covid-19 (Infections and infestations) | 6 | 3
Upper Respiratory Tract Infection (Infections and infestations) | 5 | 7
Urinary Tract Infection (Infections and infestations) | 5 | 7
Fatigue (General disorders) | 10 | 9
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 6 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 7
Nausea (Gastrointestinal disorders) | 7 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-12-05): https://cdn.clinicaltrials.gov/large-docs/99/NCT03701399/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/99/NCT03701399/SAP_001.pdf